CLINICAL TRIAL: NCT03904368
Title: The Value of Myomectomy in Women With Intramural Myoma Before IVF. A Randomized Controlled Trial
Brief Title: The Value of Myomectomy in Women With Intramural Myoma Before IVF.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55
Record Dates: First submitted 2019-03-31; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Fibroid Uterus; IVF
MeSH Terms: conditions — Leiomyoma | interventions — Gonadotropins; Chorionic Gonadotropin; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myomectomy group (Active Comparator): women with intramural myoma not reaching endometrial cavity will undergo open myomectomy followed by ovarian stimulation for in vitro fertilization 6 months after the operation
  Interventions: Procedure: Open myomectomy; Drug: Gonadotropins; Drug: Human chorionic gonadotropin; Procedure: Ovum pick up; Procedure: Embryo transfer
- Conservative group (Active Comparator): women with intramural myoma not reaching endometrial cavity will undergo ovarian stimulation for in vitro fertilization
  Interventions: Drug: Gonadotropins; Drug: Human chorionic gonadotropin; Procedure: Ovum pick up; Procedure: Embryo transfer

INTERVENTIONS:
Procedure: Open myomectomy — laparotomy then enucleation of the myoma followed by closure of the myometrial cavity
  Arms: Myomectomy group
Drug: Gonadotropins — Gonadotropin stimulation of follicular growth
  Other Names: Controlled Ovarian stimulation
Drug: Human chorionic gonadotropin — HCG triggering of ovulation
  Other Names: Ovulation triggering
Procedure: Ovum pick up — 34 to 36 hours after HCG triggering
Procedure: Embryo transfer — Transfer of 2 grade 1 embryo on day 2,3 or 5 from oocyte retrieval

SUMMARY:
Women with intramural myoma not reaching the endometrial cavity will be randomized to either open myomectomy or no intervention . The participants will be assessed through full history-taking with special consideration to age and the duration, type, and cause of infertility. The medical examination included general, abdominal, and vaginal examinations. Finally, an ultrasonography examination was performed to check for the presence of three or more preantral follicles and to exclude ovarian cysts. On day 3 of a natural cycle, a baseline levels of FSH, luteinizing hormone (LH),

, estradiol and anti-Müllerian hormone (AMH).Ovarian stimulation was performed using a long, antagonist, or short protocol. They were assigned to one of the 2 groups according to having an intramural myoma not indenting the cavity or not. All will be followed up by transvaginal ultrasonography . When two or more follicles had reached a mean diameter of 18 mm, oocyte maturation was triggered by intramuscular administration of hCG. Embryo transfer will be done at day 2, 3 or 5 according to the circumstances.

DETAILED DESCRIPTION:
Women with intramural myoma not reaching the endometrial cavity will be randomized to either open myomectomy or no intervention .The participants will be assessed through full history-taking with special consideration to age and the duration, type, and cause of infertility. The medical examination included general, abdominal, and vaginal examinations. Finally, an ultrasonography examination was performed to check for the presence of three or more preantral follicles and to exclude ovarian cysts. On day 3 of a natural cycle, a baseline levels of FSH, luteinizing hormone (LH),

, estradiol and anti-Müllerian hormone (AMH).Ovarian stimulation was performed using a long, antagonist, or short protocol. They were assigned to one of the 2 groups according to having an intramural myoma not indenting the cavity or not. All will be followed up by transvaginal ultrasonography . When two or more follicles had reached a mean diameter of 18 mm, oocyte maturation was triggered by intramuscular administration of hCG. Embryo transfer will be done at day 2, 3 or 5 according to the circumstances.

ELIGIBILITY:
Inclusion Criteria:

* • age younger than 40 years

  * FSH) less than 10 IU/L
  * serum prolactin level normal
  * uterine cavity abnormality was excluded by hysteroscopy or hysterosalpingography

Exclusion Criteria:

* abnormal endocrine function (e.g. abnormal thyroid or adrenal function)
* ovarian cysts,
* hydrosalpinx
* endometrial polyps
* male partner with azoospermia
* ICSI performed for preimplantation genetic diagnosis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  appearance of one or more intrauterine gestational sac by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided